CLINICAL TRIAL: NCT05233800
Title: Testing mHealth Delivery of Cognitive Behavioral Therapy for Insomnia to Breast Cancer Survivors
Brief Title: mHealth for Breast Cancer Survivors With Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Media Rez (Unknown)
Responsible Party: Principal Investigator, Hannah Arem, Scientific Director, Implementation Science, Medstar Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 4298
Record Dates: First submitted 2022-01-20; First posted 2022-02-10 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer Survivor; Insomnia
Keywords: Breast Cancer Survivor; Insomnia; mHealth; Digital Health; Cognitive Behavioral Therapy for Insomnia (CBT-I)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Voice-Activated Smart Speaker Program (Experimental): Faster Asleep
  Interventions: Behavioral: Faster Asleep Smart Speaker Program
- Website (Active Comparator): Faster Asleep Website
  Interventions: Behavioral: Faster Asleep Website

INTERVENTIONS:
Behavioral: Faster Asleep Smart Speaker Program — Participants will receive a smart speaker device with a pre-loaded Faster Asleep program. Participants will be asked to engage with the program daily, either using the voice-activated speakers or an accompanying smart-phone app. The study duration is six-weeks and is completed individually using fully automated interaction to deliver components of cognitive behavioral therapy for insomnia.
  Arms: Voice-Activated Smart Speaker Program
Behavioral: Faster Asleep Website — Controls will have access to a website with information about CBT-I and breast cancer survivorship and will be told to engage with the website as desired. The content will be drawn from the education script that is programmed into the phone app accompanying the smart speaker program.
  Arms: Website

SUMMARY:
The aim of this study is to determine the impact of the voice-activated smart speaker CBT-I components on insomnia symptoms among breast cancer survivors using a randomized clinical trial.

DETAILED DESCRIPTION:
This study is a Phase II SBIR to further test efficacy of a voice-activated technology to deliver components of cognitive behavioral therapy for insomnia (CBT-I) to breast cancer survivors (BCS) compared to a web-based control. Participants will be randomly assigned to the voice-activated or web-based treatment arms and will complete a 6-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to maintain a consistent dosing pattern if currently taking sleep medications or using cannabis for sleep
* Females; Age 18+
* Self-reported or documented diagnosis of breast cancer stage I-III or stage IV ECOG 0-1
* Completed curative treatment (surgery, radiation, chemotherapy) > 3 months prior to enrollment [ongoing adjuvant therapy permitted]
* Has not undergone other behavioral sleep treatment within the prior 12 months
* Score greater than or equal to 8 on the Insomnia Severity Index
* Able to understand and speak English

Exclusion Criteria:

* Diagnosed, untreated obstructive sleep apnea syndrome, narcolepsy, restless leg syndrome, periodic limb movement disorder, delayed sleep phase syndrome, central apnea
* Bi-polar disorder, schizophrenia, initiation of psychological treatment within three months, alcohol or drug abuse in the prior year (Alcohol >2 drinks/day or consuming 5+ drinks in a single day in the prior month). (Moderate ADHD, depression and anxiety will not be exclusion criteria.)
* Shift-work in the prior three months or anticipated during the study time
* Planned regular travel out of time zone (>1 hour) during the study period.
* Currently or planning to become pregnant during the study period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Arem, PhD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Cai Z, Tang Y, Liu C, Li H, Zhao G, Zhao Z, Zhang B. Cognitive behavioural therapy for insomnia in people with cancer. Cochrane Database Syst Rev. 2025 Oct 31;10(10):CD015176. doi: 10.1002/14651858.CD015176.pub2. PMID 41170811
- [Derived] Starling CM, Greenberg D, Lewin D, Shaw C, Zhou ES, Lieberman D, Chou J, Arem H. Voice-Activated Cognitive Behavioral Therapy for Insomnia: A Randomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2435011. doi: 10.1001/jamanetworkopen.2024.35011. PMID 39316400
- [Derived] Lewin D, Starling CM, Zhou ES, Greenberg D, Shaw C, Arem H. A novel voice interactive sleep log: concurrent validity with actigraphy and sleep diaries. J Clin Sleep Med. 2024 Feb 1;20(2):309-312. doi: 10.5664/jcsm.10878. PMID 37869974
- [Derived] Starling CM, Greenberg D, Zhou E, Lewin D, Morrow AS, Lieberman D, Shaw C, Arem H. Testing delivery of components of cognitive behavioral therapy for insomnia to breast cancer survivors by smart speaker: a study protocol. BMC Med Inform Decis Mak. 2022 Jun 21;22(1):163. doi: 10.1186/s12911-022-01902-w. PMID 35729605

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Voice-Activated Smart Speaker Program | Website
Started | 38 | 38
Completed | 35 | 35
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Voice-Activated Smart Speaker Program | Website | Total
Number analyzed (Participants) | 38 | 38 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.8) | 59.8 (8.7) | 61.2 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 38 | 76
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 36 | 38 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 9 | 16
  White | 28 | 25 | 53
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 38 | 38 | 76
Marital status [Count of Participants; unit: Participants]
  Single | 6 | 7 | 13
  Married or partnered | 25 | 24 | 49
  Divorced or separated | 5 | 5 | 10
  Widowed | 2 | 2 | 4
Employment [Count of Participants; unit: Participants]
  Full Time | 13 | 16 | 29
  Part time | 4 | 7 | 11
  Retired | 16 | 15 | 31
  Unemployed | 5 | 0 | 5
Education [Count of Participants; unit: Participants]
  High school/GED/Some college | 6 | 4 | 10
  College Degree | 14 | 16 | 30
  Graduate Degree | 18 | 18 | 36
TNM Cancer Stage at diagnosis [Count of Participants; unit: Participants] — This is using standardized self-reported cancer stage at diagnosis. For example, stage 0 is in situ, stage 1 is localized, stage 4 is metastatic.
  Participants
    Stage 0 | 0 | 2 | 2
    Stage 1 | 21 | 12 | 33
    Stage 2 | 12 | 17 | 29
    Stage 3 | 3 | 5 | 8
    Stage 4 | 2 | 2 | 4
BMI [Median (Inter-Quartile Range); unit: kg/m2] | 25.9 [24.1 to 29.7] | 25.6 [22.9 to 29.2] | 25.8 [23.6 to 29.2]

OUTCOME MEASURES:

1. Primary Outcome: Insomnia Symptoms
Description: Data will be collected on the Insomnia Severity Index (ISI) total score pre- and post-intervention as our primary outcome. The ISI is a seven-item questionnaire with response categories from 0-4 (total score 0-28) asking about sleep patterns and specifically characterizing insomnia over the two weeks prior. The ISI defines 'no clinically significant' insomnia as a score of 0-7, 'sub-threshold' insomnia as a score of 8-14, 'moderate severity clinical' insomnia' a scores of 15-21, and 'severe clinical' insomnia as a score of 22-28. Clinically relevant target for success is to achieve sub-threshold or better scores (≤14) among >80% of the intervention participants
Time Frame: 6 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Voice-Activated Smart Speaker Program | Website
Number analyzed (Participants) | 35 | 35
units on a scale | -8.4 (4.7) | -2.6 (3.5)
Statistical Analysis 1: Comparison: Voice-Activated Smart Speaker Program vs Website; Test type: Superiority; p < 0.05, Mixed Models Analysis; Mean Difference (Net) = 5.83, 95% CI 2-sided [3.84 to 7.81]

2. Secondary Outcome: Six Week Change in Sleep Efficiency
Description: Sleep efficiency is calculated by the total time sleeping over the total time in bed.
Time Frame: 6 weeks
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: proportion of time asleep/time in bed
Arm/Group | Voice-Activated Smart Speaker Program | Website
Number analyzed (Participants) | 35 | 35
proportion of time asleep/time in bed | 0.09 [0.07 to 0.11] | 0.05 [0.03 to 0.07]

3. Secondary Outcome: Six Week Change in Wake After Sleep Onset
Description: Amount of time awake during the night
Time Frame: 6 weeks
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Voice-Activated Smart Speaker Program | Website
Number analyzed (Participants) | 35 | 35
minutes | -18.6 [-23.9 to -13.36] | -9.1 [-14.6 to -3.63]

4. Secondary Outcome: Six Week Change in Sleep Onset Latency
Description: Time to fall asleep
Time Frame: 6 weeks
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Voice-Activated Smart Speaker Program | Website
Number analyzed (Participants) | 35 | 35
minutes | -13.79 [-18.2 to -9.33] | -5.46 [-10.1 to -0.86]

5. Secondary Outcome: Six Week Change in Total Sleep Time
Description: Total time asleep
Time Frame: 6 weeks
Population: Intent to treat
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Voice-Activated Smart Speaker Program | Website
Number analyzed (Participants) | 35 | 35
hours | 0.26 [0.06 to 0.45] | 0.27 [0.06 to 0.47]

6. Other Pre Specified Outcome: System Usability Scale
Description: A 10-item scale on general usability of technology. This provides a score of 0-100, with above 68 indicating better than average usability, where higher is better. This is a normalized score and not a percentage.
Time Frame: 6 weeks
Population: intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voice-Activated Smart Speaker Program | Website
Number analyzed (Participants) | 35 | 35
score on a scale | 72.2 (16.6) | 50.79 (15.9)

7. Other Pre Specified Outcome: End of Study Self-reported Sleep Quality
Description: 5-item Likert scale from Very Poor (5) to Very Good (1).
Time Frame: 6 weeks
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Voice-Activated Smart Speaker Program | Website
Number analyzed (Participants) | 35 | 35
score on a scale | 2.44 (0.08) | 3.03 (0.08)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Voice-Activated Smart Speaker Program | Website
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/00/NCT05233800/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-12): https://cdn.clinicaltrials.gov/large-docs/00/NCT05233800/ICF_001.pdf